CLINICAL TRIAL: NCT00697632
Title: Open-Label Dose-Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Daily Oral MGCD265 Administered Without Interruption to Subjects With Advanced Malignancies
Brief Title: Safety Study of Oral MGCD265 Administered Without Interruption to Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 265-101
Record Dates: First submitted 2008-05-14; First posted 2008-06-16 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Advanced Cancer
Keywords: MET; AXL; VEGFR; NSCLC; HNSCC (Head and neck squamous cell carcinoma); Tumor; Safety; Phase 1; Solid tumor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD265

INTERVENTIONS:
Drug: MGCD265 — Oral daily administration without interruption

SUMMARY:
In this study, MGCD265, a new anticancer drug under investigation, is given daily to patients with advanced malignancies to study its safety profile.

DETAILED DESCRIPTION:
MGCD265 belongs to a new class of drugs with anticancer potential, known as tyrosine kinase inhibitors. MGCD265 was shown to slow down the growth of human cancer cells in mice. Clinical studies are being pursued to evaluate the safety of MGCD265 in cancer patients.

In this study, MGCD265 is orally administered on a daily basis to patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Advanced metastatic or unresectable malignancy that is refractory to standard therapy and/or existing therapies are not likely to achieve clinical benefit, and/or the patient declines to receive standard treatment such as chemotherapy.
* Evaluable disease;
* Last dose of prior chemotherapy, radiation therapy, or investigational agents occurred at least 4 weeks before the start of therapy;
* Recovery from the adverse effects ≤ grade 1;
* Acceptable ECOG status 0, 1, or 2;
* Life expectancy greater than 3 months following study entry;
* Adequate laboratory values;
* For patients enrolling in the four expansion cohorts:

  * NSCLC patients must meet criteria for MET and/or Axl expression or,
  * HNSCC patients must meet criteria for MET and/or Axl expression or,
  * NSCLC patients must meet criteria for amplification of the MET gene locus, defined MET mutations, or rearrangements involving the AXL or MET gene locus or;
  * Patients with tumor types such as HNSCC, papillary renal carcinoma, gastric adenocarcinoma, and other solid tumors must meet criteria for amplification of the MET gene locus, defined MET mutations, or rearrangements involving the AXL or MET gene locus

Exclusion Criteria:

* Uncontrolled concurrent illness;
* History of cardiovascular illness;
* QTc > 470 msec (including subjects on medication);
* Left ventricular ejection fraction (LVEF) < 50%;
* Immunocompromised subjects;
* History of bone marrow transplant;
* Lung tumor lesions with increased likelihood of bleeding;
* Symptomatic or uncontrolled brain metastases;
* Unable to swallow oral medications or with pre-existing gastrointestinal disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-06; Primary Completion 2018-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year [Anticipated]

SECONDARY OUTCOMES:
Pharmacokinetics | 1 year [Anticipated]
Pharmacodynamics | 1 year [Anticipated]
Clinical response | 1 year [Anticipated]

CONTACTS AND LOCATIONS:
Locations (19):
- United States (12):
  - City of Hope, Duarte, California
  - UC Irvine Medical Center, Orange, California
  - UC San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, Alvin J. Siteman Cancer Center, St Louis, Missouri
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver Center, Vancouver, British Columbia
  - Jewish General Hospital, Montreal, Quebec
- South Korea (4):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Hosptial, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

REFERENCES:
- [Derived] Kollmannsberger C, Hurwitz H, Bazhenova L, Cho BC, Hong D, Park K, Reckamp KL, Sharma S, Der-Torossian H, Christensen JG, Faltaos D, Potvin D, Tassell V, Chao R, Shapiro GI. Phase I Study Evaluating Glesatinib (MGCD265), An Inhibitor of MET and AXL, in Patients with Non-small Cell Lung Cancer and Other Advanced Solid Tumors. Target Oncol. 2023 Jan;18(1):105-118. doi: 10.1007/s11523-022-00931-9. Epub 2022 Dec 2. PMID 36459255